CLINICAL TRIAL: NCT00299806
Title: A Multi-center, Open-label Study Assessing the Safety and Efficacy of 8 Week's Treatment of SPP100 (Aliskiren) Regimen in Patients With Severe Hypertension
Brief Title: SPP100 (Aliskiren) Regimen in Patients With Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A1304
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, rennin
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
Assessing the safety and efficacy of SPP100 (Aliskiren) regimen in patients with severe hypertension

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 80 years old
* Gender: Male or female
* Status: Outpatients
* severe hypertension

Exclusion Criteria:

* Patients with a clinically significant allergy
* Patients who have received other investigational drug
* Alcoholic patients

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic and diastolic blood pressure after 8 weeks
Average sitting systolic blood pressure/mean sitting diastolic blood is < 160/100 mmHg or blood pressure reduction from baseline is > 20/10 mmHg after 8 weeks
Average sitting diastolic blood pressure < 90 mmHg or a reduction from baseline of > 10 mmHg after 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals, Japan
Locations (1):
- Novartis Pharmaceuticals, Japan, Japan